CLINICAL TRIAL: NCT05797272
Title: Feasibility of In-utero Hematopoietic Stem Cell Transplantation as a Conjunctive Treatment During In-utero Blood Transfusion for Hemoglobin Bart's Hydrops Fetalis Syndrome in Hong Kong
Brief Title: In-utero Hematopoietic Stem Cell Transplantation for the Treatment of Fetuses With Bart's Hydrops Fetalis Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tak Yeung LEUNG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021.551-T
Record Dates: First submitted 2023-03-07; First posted 2023-04-04 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Haemoglobin Barts Hydrops
Keywords: in-utero transplantation; hematopoietic stem cell; Bart's syndrome; hydrops fetalis
MeSH Terms: conditions — Hydrops Fetalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fetuses with BHFS (Experimental): Fetuses of pregnant women confirmed with BHFS
  Interventions: Procedure: in-utero HSCT

INTERVENTIONS:
Procedure: in-utero HSCT — Pregnant women who are diagnosed to have BHFS affected fetuses and opt for continuation of pregnancy will undergo in-utero HSCT.

SUMMARY:
This is a prospective observational pilot study on pregnant women who are diagnosed to have Bart's hydrops fetalis syndrome (BHFS) affected fetuses and opt for continuation of pregnancy will be invited to consider undergoing in-utero hematopoietic stem cell transplantation under a research protocol, aiming to determine whether in-utero hematopoietic stem cell transplantation (HSCT) for fetuses with confirmed BHFS at the time of in-utero transfusion (IUT) of red blood cells could be feasible in Hong Kong. The participants will undergo bone marrow or peripheral blood stem cells harvest and an IUT combined with maternal stem cells.

DETAILED DESCRIPTION:
Alpha thalassemia major or hemoglobin BHFS is thought to be incompatible of life. A prevalence study conducted in Hong Kong showed 4.6% of the screened population are heterozygous carriers of deletional type alpha thalassemia, who would have 25% risk of conceiving fetuses with BHFS if both couple are carrier. Fetuses with BHFS often develop severe anaemia in utero, feature with cardiomegaly, high peak systolic velocity in middle cerebral artery (MCA PSV), thickened placenta, and eventually hydrops, which can lead to intrauterine fetal demise or early neonatal death; while the mother may also be at risk of maternal mirror syndrome which will cause significant morbidity and even mortality. As a result, when the foetuses are diagnosed with BHFS, most couple will terminate the pregnancy.

With the advance of technology, if the couples are both known to be alpha thalassemia carrier (alpha-alpha couples), they may consider pre-implantation genetic diagnosis. However, even though preimplantation genetic testing for monogenic disease (PGT-M) is a mature technique over the decades, it is still technically challenging, requires assisted reproductive technology even if the couple are fertile and relative costly. As a result, most of the alpha-alpha couples still conceive naturally. Prenatal ultrasonic surveillance is usually offered for the couples and prenatal diagnosis is required for genetic analysis to confirm BHFS when there is ultrasound feature of fetal anaemia.

Thus, the investigators propose this pilot study to determine whether in-utero hematopoietic stem cell transplantation for fetuses with confirmed alpha thalassemia major at the time of IUT of red blood cells could be feasible in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy before 26 weeks and 0 day of gestational age with a diagnosis of BHFS confirmed by chorionic villus sampling, amniocentesis or cordocentesis;
* The parents elected to pursue IUT and are willing to undergo subsequent IUT for the remainder of gestation.

Exclusion Criteria:

A) Fetal subjects:

* Fetuses having a second major anatomic anomaly (not related to the underlying thalassemia) that contributes a significant morbidity or mortality risk;
* Fetuses having a genetic or chromosomal abnormalities other than BHFS that contributes a significant morbidity or mortality risk;
* Echocardiogram or ultrasound findings that indicate a high risk of fetal demise after fetal intervention;
* Fetuses diagnosed with in-utero death prior to the actual intervention.

B) Maternal subjects:

* Maternal age < 18 years, mentally handicapped or severely ill;
* Maternal participants having one or more morbidities that would preclude bone marrow or peripheral blood stem cells harvest and fetal intervention including, but not limited to, bleeding disorder, maternal cardiac disease, maternal mirror syndrome, symptomatic maternal anemia, or if they develop preterm premature rupture of membranes or active preterm labor;
* Unable to understand English or Chinese to give consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 10 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of maternal complications | during pregnancy (up to week 40)
  Maternal participant tolerance of bone marrow or peripheral blood stem cells harvest with prior granulocyte colony-stimulating factor (G-CSF) administration:
  - Maternal participant tolerance defined as not requiring interventions for preterm labor, bleeding, infection or prolonged hospitalization. Any side effects or adverse outcome related to the procedure or related medications observed will be well documented.
Rate of survival of fetus | during pregnancy (up to week 40)
  Safety of in utero HSCT when performed at the same time as in utero blood transfusion for the fetal participant:
  - Safety for fetal participant defined by survival 24 hours after procedure, fetal survival till birth, neonatal survival through discharge of hospitalization and no evidence of graft versus host disease.

CONTACTS AND LOCATIONS:
Overall Officials: Tak Yeung LEUNG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong